CLINICAL TRIAL: NCT01870349
Title: Evaluation of Pro-inflammatory Mediators Around Astra Tech Dental Implant Abutments Following a Minimum of 6 Months of Clinical Function
Brief Title: A Comparison of Inflammatory Mediators Surrounding Titanium or Zirconium Implant Abutments
Status: Completed | Type: Observational
Sponsor: Christopher Barwacz (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry); University of Iowa (Other)
Responsible Party: Sponsor-Investigator, Christopher Barwacz, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 200911729
Record Dates: First submitted 2013-05-30; First posted 2013-06-06 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Peri-implantitis
Keywords: cytokines; dental implants; peri-implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Gingival crevicular fluids
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Titanium Implant Abutments: Gingival Crevicular Fluid Sampling
  Interventions: Procedure: Gingival Crevicular Fluid Sampling
- Zirconium Implant Abutments: Gingival Crevicular Fluid Sampling
  Interventions: Procedure: Gingival Crevicular Fluid Sampling

INTERVENTIONS:
Procedure: Gingival Crevicular Fluid Sampling — Gingival crevicular fluids will be sampled from single implant restorations that have been in function for at least 6 months

SUMMARY:
The purpose of this study is to determine whether there are differences in inflammatory markers and bone-mediator protein expression in the fluid surrounding implant abutments manufactured with either titanium or zirconium.

DETAILED DESCRIPTION:
The aim of this cross-sectional study is to utilize the paper strip-based peri-implant crevicular fluid (PICF) sampling technique to evaluate the influence that transmucosal abutment biomaterials of either titanium or zirconium oxide, which have been in situ for greater than six months, have in the expression of specific pro-inflammatory and bone-mediators.

Subjects who had previously undergone single-tooth implant replacement therapy are invited to participate and informed consent is obtained.

All participants receive a clinical and radiographic exam of the implant site that is sampled for PICF. Clinical and radiographic parameters such as implant mobility, presence or absence of supragingival plaque, and interproximal bone levels were assessed. Peri-apical radiographs, utilizing a paralleling technique, will be obtained from each implant fixture to evaluate the marginal bone level compared to baseline periapical radiographs made at the time of definitive prosthesis delivery. Each participant's implant site is isolated with cotton rolls, light air is applied over the site to eliminate the potential for ambient salivary contamination of the PICF sample. The implant site is sampled for 30 seconds at four distinct sites (mesio-buccal, disto-buccal, mesio-lingual, disto-lingual) by one clinician under loupe magnification. The fluid volumes collected on each strip will be quantified using the Periotron 8000 Instrument.

Cytokine, chemokine, and bone mediator quantities (pg/30 s) were determined using a commercial 22-multiplexed fluorescent bead-based immunoassay. Two specific multiplex kits are utilized (Milliplex MAP Human cytokine/Chemokine Immunoassay & Milliplex MAP Human Bone Panel 1B Immunoassay).

Biostatisticians are masked to the implant abutment biomaterial designations (masked as "A" and "B") during data analysis. Initial bivariate analysis using the Wilcoxon-Mann-Whitney (Wilcoxon Rank Sum) test will be employed to assess the difference in distribution between the two groups (titanium dioxide or zirconium oxide) for each cytokine/bone mediator and for age. The same approach is used to consider whether a gender difference was associated with a particular cytokine/bone mediator. Gender distribution in the two groups will be compared using the Fisher exact test. The Spearman rank correlation will be used to assess the possibility of a relationship with age for each cytokine. Rank-based regression models will be used to adjust for possible effects of age and gender for both cytokine and bone mediator levels.

ELIGIBILITY:
Inclusion Criteria::

* presence of a single-tooth implant-supported restoration bounded by natural teeth in stable occlusion
* pre-fabricated or computer aided design and computer aided manufactured (CAD/CAM) transmucosal abutments of either commercially-pure titanium dioxide or zirconium dioxide
* a minimum of 6 months of clinical function in situ.

Exclusion Criteria:

* subjects who are pregnant
* immunosuppressed subjects
* diabetes
* smokers
* alcohol or drug abuse
* systemic anti-inflammatory medication use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample, dental clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Levels of pro-inflammatory and bone mediators (pg/30 seconds) surrounding titanium vs. zirconium abutments | At least 6 months post crown placement
  Levels of pro-inflammatory and bone mediators

CONTACTS AND LOCATIONS:
Overall Officials: Chris A Barwacz, DDS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa College of Dentistry, Iowa City, Iowa, United States